CLINICAL TRIAL: NCT07076433
Title: Comparing the Efficacy of Core Stability Exercises and Pilates in Fibromyalgia Management: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Zaytoonah University of Jordan (Other)
Responsible Party: Principal Investigator, Hanan Hosny M Battesha, associate professor hanan hosny M Battesha, Al-Zaytoonah University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: fibromyalgia
Record Dates: First submitted 2025-07-15; First posted 2025-07-22 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Fibromyositis-Fibromyalgia Syndrome
Keywords: Core Stability Exercises; Pilates; Fibromyalgia; functional assessment
MeSH Terms: conditions — Fibromyalgia | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Stability Exercises (Experimental): Participants will engage in core stability exercises targeting the muscles of the trunk and pelvis, such as pelvic tilting, abdominal crunches, back extension, side bridges, and bird dog. These exercises will be performed twice a week for 6 weeks, with each session lasting 30 minutes. The intensity will be progressively increased based on individual tolerance.
  Interventions: Other: Core Stability Exercises
- Pilates: (Experimental): - Participants will undergo Pilates sessions that emphasize flexibility, posture, and core engagement. Pilates exercises will be performed twice a week for 6 weeks, with each session lasting 30 minutes. The focus will be on breathing, spinal alignment, and strengthening exercises that challenge flexibility and balance.
  Interventions: Other: Pilates:

INTERVENTIONS:
Other: Core Stability Exercises — Participants will engage in core stability exercises targeting the muscles of the trunk and pelvis, such as pelvic tilting, abdominal crunches, back extension, side bridges, and bird dog. These exercises will be performed twice a week for 6 weeks, with each session lasting 30 minutes. The intensity will be progressively increased based on individual tolerance.
  Arms: Core Stability Exercises
Other: Pilates: — Participants will undergo Pilates sessions that emphasize flexibility, posture, and core engagement. Pilates exercises will be performed twice a week for 6 weeks, with each session lasting 30 minutes. The focus will be on breathing, spinal alignment, and strengthening exercises that challenge flexibility and balance.
  Arms: Pilates:

SUMMARY:
Pilates and core stability exercises have emerged as potential interventions for Fibromyalgia (FM) , both targeting muscle strength, flexibility, and posture. However, existing studies have primarily relied on subjective self-report measures to assess outcomes. This study aims to employ more objective assessments, including biomechanical and functional measures, to compare the efficacy of core stability exercises and Pilates in improving symptoms of FM.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 35-65 years
* Diagnosed with fibromyalgia based on the American College of Rheumatology (ACR) 2010 criteria
* Able to walk independently
* Stable medication for at least 3 months prior to participation

Exclusion Criteria:

* Pregnant women
* History of significant orthopedic, cardiopulmonary, or neurological conditions
* Severe psychiatric disorders that interfere with participation
* Active substance abuse

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-25 (Actual)

PRIMARY OUTCOMES:
pain by Quantitative Sensory Testing | 6 weeks
  10 the best results
Functional Status: Fibromyalgia Impact Questionnaire (FIQ) | 6 weeks
  100 score tha best results

SECONDARY OUTCOMES:
Balance and Posture: Force Plate Balance Testing | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Al Zaytoonah University, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No